CLINICAL TRIAL: NCT04292392
Title: Comparison of Pain Levels and Opioid Usage in ACB + Periarticular Block vs. ACB + IPACK Block vs. ACB + IPACK + Periarticular Block in Patients Undergoing Primary TKA
Brief Title: Pain Levels and Opioid Usage in Three Nerve Block Cohorts in Primary TKA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Final protocol and ICF has not been approved by local IRB. No subjects have been enrolled. Study will not be pursued due to current COVID-19 pandemic.
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Arthur Malkani, Professor, Adult Reconstruction, Dept. of Orthopaedic Surgery, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20.0132
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Knee Arthropathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A - ACB + Periarticular Block (Experimental): Group A: patient will receive a preop ACB, followed by Intra-articular block during TKA surgery
  Interventions: Other: preop ACB, followed by Intra-articular block during TKA surgery
- B - ACB + IPACK Block (Experimental): Group B: patient will receive a preop ACB+IPACK block before TKA surgery only
  Interventions: Other: preop ACB+IPACK block
- C - ACB + IPACK + Periarticular Block (Experimental): Group C: patient will receive a preop ACB+IPACK block, followed by Intra-articular block during TKA surgery
  Interventions: Other: preop ACB+IPACK block, followed by Intra-articular block during TKA surgery

INTERVENTIONS:
Other: preop ACB, followed by Intra-articular block during TKA surgery — Preoperative ACB (adductor canal block), followed by a local anesthetic injection during surgery, which is comprised of the following agents and amounts:
  * Ropivacaine 5mg/ml (49.25ml)
  * Epinephrine 1mg/ml (0.5ml)
  * Ketorolac 30mg/ml (1ml)
  * Clonidine 0.1mg/ml (0.8ml)
  * Saline 48.45ml
  Arms: A - ACB + Periarticular Block
Other: preop ACB+IPACK block — Preoperative ACB (adductor canal block) and IPACK (Interspace between the Popliteal Artery and the Capsule of the posterior Knee) block
  Arms: B - ACB + IPACK Block
Other: preop ACB+IPACK block, followed by Intra-articular block during TKA surgery — Preoperative ACB (adductor canal block) and IPACK (Interspace between the Popliteal Artery and the Capsule of the posterior Knee) block, followed by a local anesthetic injection during surgery, which is comprised of the following agents and amounts:
  * Ropivacaine 5mg/ml (49.25ml)
  * Epinephrine 1mg/ml (0.5ml)
  * Ketorolac 30mg/ml (1ml)
  * Clonidine 0.1mg/ml (0.8ml)
  * Saline 48.45ml
  Arms: C - ACB + IPACK + Periarticular Block

SUMMARY:
The primary objective of this study is to compare effect of combined block of ACB (adductor canal block) with IPACK (Interspace between the Popliteal Artery and the Capsule of the posterior Knee) block and/or Intra-articular block in immediate postoperative and early postop rehabilitation and pain management in patients undergoing primary TKA. The secondary objective is to review both in-hospital and post-discharge pain levels and narcotic usage of primary TKAs, with a minimum 6-week postoperative follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is indicated for a primary, unilateral TKA secondary to osteoarthritis.
2. Patient age is 22-89 at time of TKA surgery.
3. Patient agrees to participate as a study subject and signs the Informed Consent and Research Authorization document.
4. Patient is able to read and speak English.

Exclusion Criteria:

1. Patient is under the age of 22 or over the age of 89.
2. Patient's primary diagnosis is not osteoarthritis (e.g. post-traumatic arthritis).
3. Patient is scheduled to undergo a bilateral TKA surgery.
4. Patient is unable to read and speak English.

Ages: 22 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
total length of hospital stay | outcome measure will be taken at 2 weeks postoperatively
  total length of hospital stay as defined by number of days from date of surgery to date of discharge
Knee Society Score | outcome measure will be taken preoperatively (4-6 weeks prior to date of surgery) and 6 weeks (± 2 weeks) postoperatively.]
  Knee Society Score as recorded preoperatively and 6 weeks (± 2 weeks) postoperatively. The score is on a scale from 0-100. A higher value represents a better outcome
WOMAC score | outcome measure will be taken preoperatively (4-6 weeks prior to date of surgery) and 6 weeks (± 2 weeks) postoperatively
  WOMAC score as recorded preoperatively and 6 weeks (± 2 weeks) postoperatively. The score is on a scale from 0-100. In contrast to the Knee Society Score, on the WOMAC a lower value represents a better outcome.
Visual Analog Scale | outcome measure will be taken 24 hours postoperatively, 48 hours postoperatively, 72 hours postoperatively, 2 weeks (± 4 days) postoperatively, and 6 weeks (± 2 weeks) postoperatively
  The Visual Analog Scale measures the patient's level of knee pain on a scale of zero to ten via what the patient expresses verbally. The Visual Analog Scale (VAS) represents the degree of pain that the patient is experiencing at the time the measure is taken. Zero represents "pain-free". A 10 would represent pain so excruciating as to warrant emergency medical assistance, or as it is described to the patient, "the worst pain imaginable". Obviously, the lower the number, the better the outcome. There is no subscale.
Amount of narcotic medication utilized | outcome measure will be taken 24 hours postoperatively, 48 hours postoperatively, 72 hours postoperatively, 2 weeks (± 4 days) postoperatively, and 6 weeks (± 2 weeks) postoperatively
  Amount of narcotic medication utilized (daily dosage measured as a Milligram Morphine Equivalent (MME) value).
Ability to rise from a chair independently | outcome measure will be taken 24 hours postoperatively, 48 hours postoperatively, 72 hours postoperatively, 2 weeks (± 4 days) postoperatively, and 6 weeks (± 2 weeks) postoperatively
  Ability to rise from a chair independently (Yes/No)
Active range-of-motion (ROM) | outcome measure will be taken 24 hours postoperatively, 48 hours postoperatively, 72 hours postoperatively, 2 weeks (± 4 days) postoperatively, and 6 weeks (± 2 weeks) postoperatively
  Active ROM (range-of-motion) as measured by a goniometer (range of 0-135 degrees)
Distance that patient is able to walk | outcome measure will be taken 24 hours postoperatively, 48 hours postoperatively, 72 hours postoperatively, 2 weeks (± 4 days) postoperatively, and 6 weeks (± 2 weeks) postoperatively
  Distance that patient is able to walk, as measured in feet
Use of an ambulatory assistive device | outcome measure will be taken 24 hours postoperatively, 48 hours postoperatively, 72 hours postoperatively, 2 weeks (± 4 days) postoperatively, 6 weeks (± 2 weeks) postoperatively
  Use of an ambulatory assistive device (Yes/No)
Incidence of postop complications | outcome measure will be taken 6 weeks (± 2 weeks) postoperatively
  Incidence of any postoperative complication that involves hospital readmission and/or a re-operation of the surgical knee.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur L Malkani, MD, Principal Investigator — University of Louisville
Locations (1):
- Jewish Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No